CLINICAL TRIAL: NCT03627936
Title: A Randomized, Open-Label, Crossover Study to Demonstrate Bioequivalence Between Lorcaserin Extended Release (XR) Tablets Manufactured in Kawashima and Lorcaserin XR Tablets Manufactured in Zofingen Under Fasted Conditions in Healthy Subjects
Brief Title: A Study to Demonstrate Bioequivalence Between Lorcaserin Extended Release (XR) Tablets Manufactured in Kawashima and Lorcaserin XR Tablets Manufactured in Zofingen in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: APD356-A001-040
Record Dates: First submitted 2018-08-07; First posted 2018-08-14 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-08

CONDITIONS: Healthy Participants
Keywords: Lorcaserin; Bioequivalence; Extended release; Tablets; Phase 1; Healthy
MeSH Terms: interventions — lorcaserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lorcaserin 20 mg manufactured at: Zofingen (A) + Kawashima (B) (Experimental): Participants will receive a single oral dose of lorcaserin 20 milligram (mg) XR tablets manufactured at Zofingen (A) after a 10-hour overnight fast on Day 1 of treatment period 1 followed by a single oral dose of lorcaserin 20 mg XR tablet manufactured at Kawashima (B) after a 10-hour overnight fast on Day 7 of treatment period 2. A washout period of 5 days will be maintained between the 2 treatment periods.
  Interventions: Drug: Lorcaserin manufactured at Zofingen; Drug: Lorcaserin manufactured at Kawashima
- Lorcaserin 20 mg manufactured at: Kawashima (B) + Zofingen (A) (Experimental): Participants will receive a single oral dose of lorcaserin 20 mg XR tablets manufactured at Kawashima (B) after a 10-hour overnight fast on Day 1 of treatment period 1 followed by a single oral dose of lorcaserin 20 mg XR tablet manufactured at Zofingen (A) after a 10-hour overnight fast on Day 7 of treatment period 2. A washout period of 5 days will be maintained between the 2 treatment periods.
  Interventions: Drug: Lorcaserin manufactured at Zofingen; Drug: Lorcaserin manufactured at Kawashima

INTERVENTIONS:
Drug: Lorcaserin manufactured at Zofingen — Lorcaserin XR tablets manufactured at Zofingen.
  Other Names: BELVIQ XR; APD356
Drug: Lorcaserin manufactured at Kawashima — Lorcaserin XR tablets manufactured at Kawashima.
  Other Names: BELVIQ XR; APD356

SUMMARY:
The purpose of this study is to demonstrate the bioequivalence between lorcaserin XR tablets manufactured in Kawashima and lorcaserin XR tablets manufactured in Zofingen.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking, healthy participants at the time of informed consent.
* Body mass index (BMI) of 18 to 30 kilogram per square meter (kg/m^2) (inclusive) at Screening.

Exclusion Criteria:

* Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks before first dosing.
* Evidence of disease that may influence the outcome of the study within 4 weeks before first dosing; eg, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism.
* History of drug or alcohol dependency or abuse within the 2 years before Screening, or those who have a positive urine drug, cotinine, or alcohol test at Screening or Baseline.
* Participants who contravene the restrictions on concomitant medications, food and beverages.
* Currently enrolled in another clinical study or used any investigational drug or device within 4 weeks preceding informed consent.
* Receipt of blood products within 4 weeks, or donation of blood within 8 weeks, or donation of plasma within 1 week of dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2018-09-02 (Actual); Study Completion 2018-09-02 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Lorcaserin | predose and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 24, 36, 48, 72, and 96 hours postdose in each treatment period; treatment period length = 4 days
Area under the concentration-time curve from zero time to time of last quantifiable concentration (AUC [0-t]) of Lorcaserin | predose and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 24, 36, 48, 72, and 96 hours postdose in each treatment period; treatment period length = 4 days
Area under the concentration-time curve from zero time extrapolated to infinite time (AUC [0-inf]) of Lorcaserin | predose and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 24, 36, 48, 72, and 96 hours postdose in each treatment period; treatment period length = 4 days
Area under the concentration-time curve from zero time to 72 hour (AUC [0-72h]) of Lorcaserin | predose and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 24, 36, 48, and 72 hours postdose in each treatment period; treatment period length = 4 days
Time to Maximum Observed Plasma Concentration (tmax) of Lorcaserin | predose and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 24, 36, 48, 72, and 96 hours postdose in each treatment period; treatment period length = 4 days
Terminal elimination phase half-life (t½) of Lorcaserin | predose and at 2, 4, 6, 8, 10, 12, 14, 16, 18, 24, 36, 48, 72, and 96 hours postdose in each treatment period; treatment period length = 4 days

SECONDARY OUTCOMES:
Number of Participants With One or More Treatment-emergent Adverse Event (TEAE) and Serious Adverse Event (SAE) | Baseline up to 28 days after last dose of study drug (Day 35)
Number of Participants With Markedly Abnormal Laboratory Values | Baseline up to Day 11
Number of Participants With Change From Baseline in Vital Signs Parameters | Baseline, Day 1, Day 2, Day 6, Day 7, Day 8, and Day 11
Number of Participants With Clinically Significant Findings in Physical examinations | Baseline and Day 11

CONTACTS AND LOCATIONS:
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States